CLINICAL TRIAL: NCT04703465
Title: Effectiveness and Safety of Tenofovir Alafenamide for HBV Prophylaxis in HBV Negative Recipients Received Orthotopic Liver Transplant With HBcAb+ Donors
Brief Title: Tenofovir Alafenamide for HBV Prophylaxis in HBV(-) Liver Transplant Recipients With HBcAb+ Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: In the application
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: HBV; Liver Transplant Disorder
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tenofovir alafenamide (Experimental): tenofovir alafenamide 25mg daily for 48 weeks
  Interventions: Drug: Tenofovir Alafenamide 25 MG

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG — Tenofovir Alafenamide 25mg for 48 weeks will be delivered
  Other Names: Vemlidy

SUMMARY:
Liver transplantation is currently the only effective way to treat end-stage liver disease.The shortage of donor liver is still the major problem. Incidence of HBcAb+ varies between different regions. The HBcAb positive rate could be as high as 52% in China.HBcAb positive donor liver may enlarge donor pool and thus save ESLD patients. However, the use of HBcAb positive donor liver may induce HBV infection in hepatitis B negative recipient after liver transplantation. Tenofovir alafenamide (TAF) has better stability in plasma and higher liver targeting property in comparison with tenofovir (TDF), with an extra amide bond, which allows strong antiviral effect with much less doses and reducing the renal and bone injury. Our study intends to evaluate the efficacy and safety of HBV prophylaxis treatment of TAF in HBV negative patients after receiving HBcAb positive donor livers.

DETAILED DESCRIPTION:
We intent to enroll 30 patients who are HBV negative but received HBcAb+ liver. Antiviral treatment with TAF(25mg/d,oral) will be started on the first day after liver transplantation. Post-operative HBV infection is defined with positive HBV marker (HBsAg) and/or positive HBV DNA after liver transplantation. Primary outcome will be evaluated at 48 weeks. All the patients will be followed up for another at least 1 year to evaluate the long term efficacy and safety of TAF.

The primary endpoint is to calculate de novo HBV infection after liver transplantation when treating with TAF. Secondary endpoint is to evaluate the renal safety of TAF after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with written informed consent.
2. Age ≥12 years old
3. HBV negative recipients (HBV DNA undetectable and HBsAg negative) receiving HBsAg-, HBcAb+ donor liver

Exclusion Criteria:

1. Patients underwent liver re-transplantation
2. CKD (CrCl<30 ml/min by MDRD formula)
3. HBV/HCV-related OLT
4. Other solid organs transplant recipients
5. HIV coinfection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
De novo HBV infected rate after liver transplantation at 48 weeks | 48 weeks
  Primary outcome is to calculate de novo HBV infection after liver transplantation when treating with TAF.

SECONDARY OUTCOMES:
48 weeks Renal safety of TAF after liver transplantation. | 48 weeks
  Secondary outcome is to evaluate changes in renal function (Serum Creatinine, eGFR, β2-MG: Cr, RBP:Cr) at 48 weeks.
96 weeks Renal safety of TAF after liver transplantation. | 96 weeks
  Secondary outcome is to evaluate changes in renal function (Serum Creatinine, eGFR, β2-MG: Cr, RBP:Cr) at 96 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, MD., Ph.D., Study Chair — RenJi Hospital; Zhifeng Xi, MD., Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No